CLINICAL TRIAL: NCT07115732
Title: A Prospective Single Centre Post Market Clinical Follow-up Study of the JRI Orthopaedic ACE Acetabular Cup System in Spain
Brief Title: ACE Acetabular Cup Spanish PMCF Study
Status: Not yet recruiting | Type: Observational
Sponsor: JRI Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: JRI-CS-011
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hip Disease
Keywords: Total Hip Replacement; Patient reported outcome measures; Post Market Clinical Follow-up / Post Market Surveillance
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ACE Acetabular Cup System with XLPE Liner
  Interventions: Device: Total Hip Replacement
- ACE Acetabular Cup System with Ceramic Liner
  Interventions: Device: Total Hip Replacement

INTERVENTIONS:
Device: Total Hip Replacement — Primary elective total hip replacement

SUMMARY:
A total hip replacement is one of the most successful and cost-effective surgical procedures in orthopaedics, involving the replacement of both the hip ball and socket. Its goal is to provide pain relief and enable the patient to return to a normal lifestyle. JRI Orthopaedics have developed the ACE Acetabular Cup System, which has an H-A.C. coating to promote osseointegration of the device within the host bone. To increase the surgeon's choice and thus suitability for the patient, there is the option of three different socket liners (ceramic, polymer, or dual mobility).

To ensure maximum safety and performance of medical devices, surveillance of the device should be carried out over the device's lifetime. This study is a 10-year surveillance study to assess the clinical, functional, and radiological outcomes of the CE-marked ACE Acetabular Cup System. This will be done by examining patient outcomes through questionnaires, reviews of X-rays, and recording any complications in patients who have received a total hip replacement using the ACE Acetabular Cup System at participating sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed suitable for elective primary THR, as per indications in the IFU.
* Male or female, 18 years to 85 years.

Exclusion Criteria:

* Patients who are unable to provide written informed consent.
* Patients deemed unsuitable for THR, as per contra-indications in the IFU.
* Patients indicated for THR as a result of trauma (i.e. neck of femur fracture).
* Patients who are pregnant (exclusion criteria for THR in general).
* Patients receiving implants other than the approved combination, i.e. an ACE Acetabular Cup System with a JRI femoral stem and head.
* Patients who are unable to comply with the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require elective primary total hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip Score | 3 years post-op
  A patient completed functional score to assess pain and function of the affected hip joint. Score range: 0 (worse) to 48 (best)

SECONDARY OUTCOMES:
Implant Survivorship | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  Implant survivorship based on revision rate and determined using the Kaplan-Meier analysis method
Oxford Hip Score | 6 months, 1 year, 5 years, 7 years and 10 years post-op
  A patient completed functional score to assess pain and function of the affected hip joint. Score range: 0 (worse) to 48 (best)
Modified Harris Hip Score | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  A patient completed functional score to assess pain and function of the affected hip joint. Score range: 0 (worse) to 100 (best)
EQ-5D-5L | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  A patient completed functional score to assess quality of life of the patient. Score range: -0.594 (worse) to 1.0 (best).
Radiological Assessment | 1 year, 5 years and 10 years post-op
  Radiographs reviewed for signs of radiolucencies, osteolysis, sclerosis and atrophy around the device

OTHER OUTCOMES:
Adverse Device Effects | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  Trends and anaylsis or adverse device effects reported

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Granollers, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No